CLINICAL TRIAL: NCT01458210
Title: Effect of Dulaglutide (LY2189265) on Oral Contraceptive Pharmacokinetics in Healthy Female Subjects
Brief Title: A Study of the Effect of Dulaglutide on How the Body Handles Oral Contraceptive in Healthy Female Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11555; H9X-MC-GBCQ (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-10-19; First posted 2011-10-24 (Estimated); Results first posted 2014-10-08 (Estimated); Last update posted 2014-10-08 (Estimated); Status verified 2014-10

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Moxifloxacin; dulaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ortho-Cyclen (OC) Alone (Period 1); OC+Dulaglutide (Period 2) (Experimental): Ortho-Cyclen (OC) (0.25 milligram [mg] norelgestromin [NGMN] + 0.035 mg ethinyl estradiol [EE] [active tablets] for 21 days + non-active tablets for 7 days): A 28-day course of OC consists of 0.25 mg NGMN and 0.035 mg EE (active tablets), administered orally, once per day for 21 days, then non-active tablets, administered orally, once per day for 7 days. Participants received the first 28-day course (Lead-in) followed by 2 subsequent 28-day courses (Periods 1 and 2, respectively). Following the Lead-in period, the Period 1 sample was taken during the first 28-day course and the Period 2 sample was taken during the second 28-day course.
  Dulaglutide: A single, 1.5-mg subcutaneous injection on Day 19 of Period 2.
  Interventions: Drug: Ortho-Cyclen; Biological: Dulaglutide

INTERVENTIONS:
Drug: Ortho-Cyclen — Administered orally
Biological: Dulaglutide — Administered subcutaneously
  Other Names: LY2189265

SUMMARY:
The purpose of this study is to look at how the body processes oral contraceptive (OC), using Ortho-Cyclen, as a commonly prescribed combination oral contraceptive in healthy female participants, and the effect of dulaglutide on how Ortho-Cyclen is processed by the body. Information about any side effects that may occur will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Are females of child-bearing potential, and who are overtly healthy as determined by medical history and physical examination

  * As it is possible that dulaglutide may cause the oral contraceptive (OC) tablet to be less effective than usual, participants will be required to use 2 additional highly effective methods of contraception from the screening appointment until 2 months after the poststudy follow-up appointment. Additional methods of contraception may include the following: a non-hormonal intrauterine device with spermicide; male or female condom with spermicide; contraceptive sponge with spermicide; diaphragm with spermicide; cervical cap with spermicide; sterile sexual partner; or abstinence (participants reporting abstinence who become sexually active while on the study must agree to use other additional methods of contraception). The pregnancy test result must be negative at screening and at each check-in
* Have a body mass index (BMI) of between 18.5 and 30.0 kilogram-meter squared (kg/m^2), at screening
* Have no clinically significant findings, as determined by the investigator, upon bimanual pelvic and breast examinations, at screening (provision of previous gynecological examination documentation may be accepted)
* Have clinical laboratory test results within the normal reference range for the population or investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator
* Have venous access sufficient to allow for blood sampling
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures and restrictions
* Have given written informed consent approved by Lilly and the ethical review board (ERB) governing the site

Exclusion Criteria:

* Are currently enrolled in, have completed or discontinued within the last 30 days from, a clinical trial involving an investigational product, or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Have known allergies to Ortho-Cyclen, dulaglutide, or to related compounds or to any components of either formulation
* Are persons who have previously completed or withdrawn from this study or any other study investigating dulaglutide within 3 months prior to screening or have received glucagon-like peptides or incretin mimetics in the 3 months prior to screening
* Have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study
* Have an abnormal blood pressure (BP) (after at least 5 minutes sitting) that, in the opinion of the investigator, increases the risks associated with participating in the study
* Have a history or presence of respiratory, hepatic, renal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data
* Have a history or presence of cardiovascular disorder (including myocardial infarction, cerebrovascular accident, coronary artery disease, venous thromboembolism, arrhythmia [judged by the investigator to be clinically significant], or angina) within the last year, have symptoms or signs of congestive heart failure, or are expected to require coronary artery bypass surgery or angioplasty
* Have a history or presence of pancreatitis (history of chronic pancreatitis or idiopathic acute pancreatitis) or gastrointestinal disorder, for example relevant esophageal reflux or gall bladder disease, or any gastrointestinal disease which impacts gastric emptying (GE) (such as, gastric bypass surgery, pyloric stenosis, with the exception of appendectomy) or could be aggravated by glucagon-like-peptide 1 (GLP-1) analogs. Participants with dyslipidemia, and participants who had cholecystolithiasis (removal of gall stones) and/or cholecystectomy (removal of gall bladder) in the past, with no further sequelae, may be included in the study at the discretion of the screening physician
* Show evidence of significant active neuropsychiatric disease
* Have family history of medullary thyroid cancer (MTC) or a genetic condition that predisposes to MTC
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening
* Show evidence of human immunodeficiency virus (HIV) infection and/or positive HIV antibodies
* Show evidence of hepatitis C and/or positive hepatitis C antibody
* Show evidence of hepatitis B and/or positive hepatitis B surface antigen
* Are women with a positive pregnancy test or women who are lactating
* Have used or intend to use St John's Wort within 21 days of study drug administration or are unable/unwilling to adhere to the study drug restrictions
* Have donated blood of more than 500 milliliter (mL) within the last month prior to admission of the lead-in phase
* Have an average weekly alcohol intake that exceeds 14 units per week, or are unwilling to stop alcohol consumption for 48 hours prior to each admission to the clinical research unit (CRU) and while resident at the CRU (1 unit = 12 ounce [oz] or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits)
* Use of any tobacco- or nicotine-containing products (including but not limited to cigarettes, pipes, cigars, chewing tobacco, nicotine patches, nicotine lozenges, or nicotine gum) within 6 months prior to admission into the lead-in phase
* Have taken injectable contraceptives or have used hormonal implants within 12 months of enrollment to this study or topical controlled delivery contraceptives (patch) or hormonal intrauterine devices (such as, Mirena® device) within 3 months prior to enrollment of this study
* The history or presence of any contraindications to the combined OC tablet including thrombosis and a history of thromboembolic disease, recurrent jaundice, acute or chronic liver disease, migraines, undiagnosed vaginal bleeding, significant hyperlipidemia, hepatic adenoma, and mammary, endometrial, or hepatic carcinoma or any other estrogen-dependent neoplasia (known or suspected)
* In the opinion of the investigator or sponsor, are unsuitable for inclusion in the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2011-10; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas, United States

REFERENCES:
- [Derived] de la Pena A, Cui X, Geiser J, Loghin C. No Dose Adjustment is Recommended for Digoxin, Warfarin, Atorvastatin or a Combination Oral Contraceptive When Coadministered with Dulaglutide. Clin Pharmacokinet. 2017 Nov;56(11):1415-1427. doi: 10.1007/s40262-017-0531-7. PMID 28357715

RESULTS

PARTICIPANT FLOW:
Groups:
- Overall Study: Ortho-Cyclen (OC) (0.25 milligram [mg] norelgestromin [NGMN] + 0.035 mg ethinyl estradiol [EE] [active tablets] for 21 days + non-active tablets for 7 days): A 28-day course of OC consists of 0.25 mg NGMN and 0.035 mg EE (active tablets), administered orally, once per day for 21 days, then non-active tablets, administered orally, once per day for 7 days. Participants received the first 28-day course (Lead-in) followed by 2 subsequent 28-day courses (Periods 1 and 2, respectively).
  Dulaglutide: A single, 1.5-mg subcutaneous injection on Day 19 of Period 2.
Period: Lead-in (1st Course of Ortho-Cyclen)
Arm/Group | Overall Study
Started | 22
Received at Least One Dose of Study Drug | 22
Completed | 22
Not Completed | 0
Period: Ortho-Cyclen Alone (Period 1)
Arm/Group | Overall Study
Started | 22
Completed | 18
Not Completed | 4
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 2
Period: Ortho-Cyclen + Dulaglutide (Period 2)
Arm/Group | Overall Study
Started | 18 (1 participant received Ortho-Cyclen, discontinued due to Adverse Event before receiving Dulaglutide.)
Completed | 15
Not Completed | 3
Not completed — Withdrawal by Subject | 2
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Participants who received at least 1 dose of study drug.
Arm/Group | Overall Study
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.4 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Area Under the Concentration Versus Time Curve (AUC) at Steady State of Ortho-Cyclen - Norelgestromin (NGMN)
Time Frame: Day 21 during Periods 1 and 2: Pre-dose and up to 24 hours post-dose
Population: Participants who received at least 1 dose of study drug with evaluable norelgestromin (NGMN) concentration data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picograms*hour/milliliter (pg*h/mL)
Groups:
- Ortho-Cyclen Alone (Period 1): Ortho-Cyclen (OC) (0.25 milligram [mg] norelgestromin [NGMN] + 0.035 mg ethinyl estradiol [EE] [active tablets] for 21 days + non-active tablets for 7 days): A 28-day course of OC consists of 0.25 mg NGMN and 0.035 mg EE (active tablets), administered orally, once per day for 21 days, then non-active tablets, administered orally, once per day for 7 days. Participants received the first 28-day course (Lead-in) followed by 2 subsequent 28-day courses (Periods 1 and 2, respectively). Following the Lead-in period, the Period 1 sample was taken during the first 28-day course.
- Ortho-Cyclen + Dulaglutide (Period 2): Ortho-Cyclen (OC) (0.25 milligram [mg] norelgestromin [NGMN] + 0.035 mg ethinyl estradiol [EE] [active tablets] for 21 days + non-active tablets for 7 days): A 28-day course of OC consists of 0.25 mg NGMN and 0.035 mg EE (active tablets), administered orally, once per day for 21 days, then non-active tablets, administered orally, once per day for 7 days. Participants received the first 28-day course (Lead-in) followed by 2 subsequent 28-day courses (Periods 1 and 2, respectively). Following the Lead-in period, the Period 2 sample was taken during the second 28-day course.
  Dulaglutide: A single, 1.5-mg subcutaneous injection on Day 19 of Period 2.
Arm/Group | Ortho-Cyclen Alone (Period 1) | Ortho-Cyclen + Dulaglutide (Period 2)
Number analyzed (Participants) | 19 | 14
picograms*hour/milliliter (pg*h/mL) | 17900 (26) | 16000 (18)

2. Primary Outcome: Pharmacokinetics: Maximum Observed Drug Concentration (Cmax) of Ortho-Cyclen - Norelgestromin (NGMN)
Time Frame: Day 21 during Periods 1 and 2: Pre-dose and up to 24 hours post-dose
Population: Participants who received at least 1 dose of study drug with evaluable norelgestromin (NGMN) concentration data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picograms per milliliter (pg/mL)
Arm/Group | Ortho-Cyclen Alone (Period 1) | Ortho-Cyclen + Dulaglutide (Period 2)
Number analyzed (Participants) | 19 | 14
picograms per milliliter (pg/mL) | 1770 (24) | 1310 (30)

3. Primary Outcome: Pharmacokinetics: Time of Maximum Observed Drug Concentration (Tmax) of Ortho-Cyclen - Norelgestromin (NGMN)
Time Frame: Day 21 Periods 1 and 2: Pre-dose and up to 24 hours post-dose
Population: Participants who received at least 1 dose of study drug with evaluable norelgestromin (NGMN) concentration data.
Measure: Median (Full Range); unit: hours
Arm/Group | Ortho-Cyclen Alone (Period 1) | Ortho-Cyclen + Dulaglutide (Period 2)
Number analyzed (Participants) | 19 | 14
hours | 3.00 [1.00 to 4.00] | 4.00 [1.50 to 6.00]

4. Primary Outcome: Pharmacokinetics: Area Under the Concentration Versus Time Curve (AUC) at Steady State of Ortho-Cyclen - Ethinyl Estradiol (EE)
Time Frame: Day 21 during Periods 1 and 2: Pre-dose and up to 24 hours post-dose
Population: Participants who received at least 1 dose of study drug with evaluable ethinyl estradiol (EE) concentration data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picograms*hour/milliliter (pg*h/mL)
Arm/Group | Ortho-Cyclen Alone (Period 1) | Ortho-Cyclen + Dulaglutide (Period 2)
Number analyzed (Participants) | 19 | 14
picograms*hour/milliliter (pg*h/mL) | 901 (23) | 903 (28)

5. Primary Outcome: Pharmacokinetics: Maximum Observed Drug Concentration (Cmax) of Ortho-Cyclen - Ethinyl Estradiol (EE)
Time Frame: Day 21 during Periods 1 and 2: Pre-dose and up to 24 hours post-dose
Population: Participants who received at least 1 dose of study drug with evaluable ethinyl estradiol (EE) concentration data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picograms per milliliter (pg/mL)
Arm/Group | Ortho-Cyclen Alone (Period 1) | Ortho-Cyclen + Dulaglutide (Period 2)
Number analyzed (Participants) | 19 | 14
picograms per milliliter (pg/mL) | 86.9 (22) | 76.2 (34)

6. Primary Outcome: Pharmacokinetics: Time of Maximum Observed Drug Concentration (Tmax) of Ortho-Cyclen - Ethinyl Estradiol (EE)
Time Frame: Day 21 during Periods 1 and 2: Pre-dose and up to 24 hours post-dose
Population: Participants who received at least 1 dose of study drug with evaluable ethinyl estradiol (EE) concentration data.
Measure: Median (Full Range); unit: hours
Arm/Group | Ortho-Cyclen Alone (Period 1) | Ortho-Cyclen + Dulaglutide (Period 2)
Number analyzed (Participants) | 19 | 14
hours | 3.00 [1.00 to 4.00] | 4.00 [1.50 to 6.00]

ADVERSE EVENTS:
Time Frame: Ortho-Cyclen alone includes Period 1 and Day 1 through Day 18 (before the administration of dulaglutide) in Period 2. Ortho-Cyclen + Dulaglutide includes from Day 19 (postdose of dulaglutide) in Period 2 through the end of the study.
Groups:
- Lead-in (1st Course of Ortho-Cyclen): Ortho-Cyclen (OC) (0.25 milligram [mg] norelgestromin [NGMN] + 0.035 mg ethinyl estradiol [EE] [active tablets] for 21 days + non-active tablets for 7 days): A 28-day course of OC consists of 0.25 mg NGMN and 0.035 mg EE (active tablets), administered orally, once per day for 21 days, then non-active tablets, administered orally, once per day for 7 days. Participants received the first 28-day course (Lead-in).
- Ortho-Cyclen Alone: Ortho-Cyclen (OC) (0.25 milligram [mg] norelgestromin [NGMN] + 0.035 mg ethinyl estradiol [EE] [active tablets] for 21 days + non-active tablets for 7 days): A 28-day course of OC consists of 0.25 mg NGMN and 0.035 mg EE (active tablets), administered orally, once per day for 21 days, then non-active tablets, administered orally, once per day for 7 days. Participants received the first 28-day course (Lead-in) followed by 2 subsequent 28-day courses (Periods 1 and 2, respectively).
- Ortho-Cyclen + Dulaglutide: Ortho-Cyclen (OC) (0.25 milligram [mg] norelgestromin [NGMN] + 0.035 mg ethinyl estradiol [EE] [active tablets] for 21 days + non-active tablets for 7 days): A 28-day course of OC consists of 0.25 mg NGMN and 0.035 mg EE (active tablets), administered orally, once per day for 21 days, then non-active tablets, administered orally, once per day for 7 days. Participants received the first 28-day course (Lead-in) followed by 2 subsequent 28-day courses (Periods 1 and 2, respectively).
  Dulaglutide: A single, 1.5-mg subcutaneous injection on Day 19 of Period 2.
Arm/Group | Lead-in (1st Course of Ortho-Cyclen) | Ortho-Cyclen Alone | Ortho-Cyclen + Dulaglutide
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/17
Other Adverse Events (participants affected / at risk) | 5/22 | 14/22 | 11/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lead-in (1st Course of Ortho-Cyclen) (N=22) | Ortho-Cyclen Alone (N=22) | Ortho-Cyclen + Dulaglutide (N=17)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 2 (2)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 7 (7)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 6 (14)
Asthenia (General disorders) | 1 (1) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 8 (10) | 7 (7)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 1 (1) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (7) | 1 (1)
Peripheral coldness (Vascular disorders) | 0 (0) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days